CLINICAL TRIAL: NCT02628990
Title: The Effect of Plant Stanol Ester Yoghurt Drinks With or Without Added Camelina Oil on Serum Lipids in Comparison to Placebo in Subjects With Mildly to Moderately Elevated Serum Cholesterol Concentrations
Brief Title: Lipid-lowering Effect of Plant Stanol Ester Yoghurt Drinks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Raisio Group (Industry)
Collaborators: University of Turku (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YD2005
Record Dates: First submitted 2015-12-01; First posted 2015-12-11 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Hypercholesterolemia; Hyperlipidemias; Dyslipidemias
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias; Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1.6 g plant stanols (Experimental): A yoghurt drink containing plant stanol ester (1.6 grams plant stanols), consumed with a meal daily for 4 weeks
  Interventions: Other: 1.6 g plant stanols
- 2 g plant stanols (Experimental): A yoghurt drink containing plant stanol ester (2 grams plant stanols), consumed with a meal daily for 4 weeks
  Interventions: Other: 2 g plant stanols
- 1.6 g plant stanols and camelina oil (Experimental): A yoghurt drink containing plant stanol ester (1.6 grams plant stanols) and camelina oil (2 g), consumed with a meal daily for 4 weeks
  Interventions: Other: 1.6 g plant stanols and camelina oil
- 2 g plant stanols and camelina oil (Experimental): A yoghurt drink containing plant stanol ester (2 grams plant stanols) and camelina oil (2 g), consumed with a meal daily for 4 weeks
  Interventions: Other: 2 g plant stanols and camelina oil
- Placebo (Placebo Comparator): A placebo yoghurt drink, consumed with a meal daily for 4 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Other: 1.6 g plant stanols — Lipid-lowering effect of Yoghurt Drink with 1.6 g plant stanols
  Arms: 1.6 g plant stanols
Other: 2 g plant stanols — Lipid-lowering effect of Yoghurt Drink with 2 g plant stanols
  Arms: 2 g plant stanols
Other: 1.6 g plant stanols and camelina oil — Lipid-lowering effect of Yoghurt Drink with 1.6 g plant stanols and camelina oil
  Arms: 1.6 g plant stanols and camelina oil
Other: 2 g plant stanols and camelina oil — Lipid-lowering effect of Yoghurt Drink with 2 g plant stanols and camelina oil
  Arms: 2 g plant stanols and camelina oil
Other: Placebo — Lipid-lowering effect of Placebo Yoghurt Drink
  Arms: Placebo

SUMMARY:
The aim is to investigate the effects of yoghurt drinks containing two doses of plant stanol ester either with or without added camelina oil on the serum cholesterol levels in moderately hypercholesterolemic subjects

ELIGIBILITY:
Inclusion Criteria:

* BMI < 30 kg/m2
* moderate hypercholesterolemia (fasting total cholesterol between 5-8 mmol/l)
* serum triglycerides < 3 mmol/l.
* normal liver, kidney and thyroid function
* subjects must voluntarily sign the informed consent

Exclusion Criteria:

* use of cholesterol lowering foods or dietary supplements within 21 days before the start of the intervention
* lipid lowering medication
* history of unstable coronary artery disease (myocardial infarction, coronary artery bypass craft (CABG), percutaneous transluminal coronary angioplasty (PTCA) within the previous 6 months, diabetes, hyperglycemia, temporal ischemic attack and malignant diseases
* pregnancy or lactation
* alcohol abuse
* subjects with intolerance to any ingredient of the test products

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2005-06; Primary Completion 2005-08 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Percentual change in serum LDL-cholesterol | 4 weeks
  Percentual change [end of intervention - start of intervention] in serum LDL-cholesterol between experimental and placebo groups
Absolute change in serum LDL-cholesterol | 4 weeks
  Absolute change [end of intervention - start of intervention] in serum LDL-cholesterol between experimental and placebo groups, mmol/l

SECONDARY OUTCOMES:
Percentual change in serum total cholesterol | 4 weeks
  Percentual change [end of intervention - start of intervention] in serum total cholesterol between experimental and placebo groups
Absolute change in serum total cholesterol | 4 weeks
  Absolute change [end of intervention - start of intervention] in serum total cholesterol between experimental and placebo groups, mmol/l
Percentual change in serum non-HDL cholesterol | 4 weeks
  Percentual change [end of intervention - start of intervention] in serum nonHDL cholesterol between experimental and placebo groups
Absolute change in serum non-HDL cholesterol | 4 weeks
  Absolute change [end of intervention - start of intervention] in serum nonHDL cholesterol between experimental and placebo groups, mmol/l
Percentual change in serum triglycerides | 4 weeks
  Percentual change [end of intervention - start of intervention] in serum triglycerides between experimental and placebo groups
Absolute change in serum triglycerides | 4 weeks
  Absolute change [end of intervention - start of intervention] in serum triglycerides between experimental and placebo groups, mmol/l

REFERENCES:
- [Derived] Salo P, Kuusisto P. Cholesterol Lowering Effect of Plant Stanol Ester Yoghurt Drinks with Added Camelina Oil. Cholesterol. 2016;2016:5349389. doi: 10.1155/2016/5349389. Epub 2016 Feb 21. PMID 26998355